CLINICAL TRIAL: NCT00209885
Title: Optimal Multimodal Analgesia in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMA-LC01
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Cholecystolithiasis
MeSH Terms: conditions — Cholecystolithiasis | interventions — Gabapentin; Esketamine; Lidocaine; Droperidol

INTERVENTIONS:
Drug: Gabapentin
Drug: S-ketamine
Drug: Lidocaine
Drug: Droperidol

SUMMARY:
To test the current standard of care (SOC) treatment for laparoscopic cholecystectomy with a group receiving SOC + additional perioperative analgesics in terms of postoperative abilities, PONV, pain and discharge time from the PACU

DETAILED DESCRIPTION:
Aim of the study: to compare postoperative complaints (PONV, pain, etc) and PACU discharge time between two groups:

* A: standard of care (SOC)receiving intraoperative dexamethasone, ondansetron, ketorolac, and general anaesthesia with propofol, remifentanil and cisatracurium
* B: SOC + preoperative gabapentin, intraoperative lidocain infusion, s-ketamin and droperidol.

Primary endpoints:

* postoperative abilities over time
* discharge time from PACU according to fixed criteria
* consumption of analgesics and antiemetics in the PACU

Secondary endpoints:

* degree of nursing requirements at the PACU
* General tolerability of the regimes

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic cholecystectomy
* Age above 18 years
* Written informed consent
* ASA class I-III

Exclusion Criteria:

* Planned abdominal cholecystectomy
* Intraoperative conversion of laparoscopic to laparotomic cholecystectomy
* Allergy to part of the treatment regimens
* Previous reactions to opioids (nausea, cognition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-10

PRIMARY OUTCOMES:
1. postoperative abilities over time in PACU
2. discharge time from PACU according to fixed criteria
3. consumption of analgesics and antiemetics in the PACU

SECONDARY OUTCOMES:
1. Degree of nursing requirements in the PACU
2. General tolerability of the regimens

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Jensen, M.D., Principal Investigator — Dept of Anaesthesia, Acute Pain Service, Hvidovre Hospital, Copenhagen, Denmark; Claus Lund, dr.med.sci, Study Chair — Dept of Anaesthesia, Hvidovre Hospital, Copenhagen, Denmark
Locations (1):
- Dept of Anaesthesia, Hvidovre Hospital, Copenhagen, Hvidovre, Denmark

REFERENCES:
- See also: URL looking into anaesthesia and surgery for cholecystectomy — http://www.postoppain.org